CLINICAL TRIAL: NCT06703320
Title: Brain Activation Pattern Caused by Immersive Virtual Reality Pathfinding Task in Stroke Patients: a Functional Near-infrared Spectroscopy Study
Brief Title: Brain Activation Pattern Caused by Immersive Virtual Reality Pathfinding Task in Stroke Patients: an FNIRS Study
Status: Recruiting | Type: Observational
Sponsor: Dingqun Bai (Other)
Responsible Party: Sponsor-Investigator, Dingqun Bai, Director of rehabilitation Medicine, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 20241122
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Cognitive Decline
Keywords: stroke; virtual reality; cognitive impairment; fNIRS
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy subjects: Healthy subjects without history of stroke or cognitive impairment.
- PSCI: Healthy subjects without history of stroke or cognitive impairment.
- NPSCI: Stroke patients without post-stroke cognitive impairment.

SUMMARY:
This is an fNIRS study performed to investigate Brain Activation Pattern Caused by Immersive Virtual Reality Pathfinding Task in Stroke Patients.

DETAILED DESCRIPTION:
This was an initial screening and preliminary intervention study. Both healthy subject and stroke patients will be included in this study. Brain functional activation of each subject during Immersive Virtual Reality Pathfinding Task will be evaluated using functional near-infrared spectroscopy (fNIRS). Cognitive function related scale assessment included Mental State Examination Scale (MMSE), Montreal Cognitive Assessment (MoCA), drawing clock test (DCT), Shape trials test A.B (STT-A, STT-B), standardized digital modal test (SDMT), auditory verbal learning test-Huashan version (AVLT-H), and activity of daily living (ADL) scale will be used to evaluate the function of each patient. Brain Activation Pattern Caused by Immersive Virtual Reality Pathfinding Task will be identified by by comparing differences in brain activation and brain network connectivity between patients and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Stroke patients:

1. Diagnosis of stroke confirmed by neuroimaging (CT or MRI)
2. 18-80 years old
3. Able to complete the cognitive task
4. Able to follow instructions to complete the trial
5. Patients who signed an informed consent form.

Healthy Subjects:

1. No abnormalities on cranial
2. 18-80 years old
3. Able to complete cognitive task
4. Able to follow instructions to complete the trial
5. not taking medications.
6. Subjects who signed an informed consent form.

Exclusion Criteria:

Stroke patients:

1. Inability to tolerate the test due to organic diseases
2. Serious mental illness that prevents them from cooperating with or tolerating the trial
3. Pregnant or lactating women
4. Had metal implants, a history of other neurological disorders, acute cardiopulmonary dysfunction.

Healthy Subjects:

1. Inability to tolerate the test due to organic diseases
2. Serious mental illness that prevents them from cooperating with or tolerating the trial.
3. Pregnant or lactating women
4. Had metal implants, a history of other neurological disorders, acute cardiopulmonary dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with stroke in the inpatient ward of the Department of Rehabilitation Medicine, The First Affiliated Hospital of Chongqing Medical University.
  Healthy subjects recruited through the Department of Rehabilitation Medicine, The First Affiliated Hospital of Chongqing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Brain Activation Pattern Caused by Immersive Virtual Reality Pathfinding Task in Stroke Patients | 1 day
  Comparison of differences in brain activation [HbO2 (mmol/L*mm)] between patients with post-stroke cognitive impairment and patients without post-stroke cognitive impairment or healthy subjects during Immersive Virtual Reality Pathfinding Task.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, the First Affiliated Hospital of Chongqing Medical University, Chongqing,, Chongqing, Chongqing 400010, Chongqing, Chongqing Municipality, China